CLINICAL TRIAL: NCT01980524
Title: HYPOglycemia Linked to Cardiac sTEatoSIS? - Identifying Mechanisms That Explain Adverse Cardiovascular Outcome Associated With Intensive Glucose Control in Patients With Diabetes (HYPOTESIS)
Brief Title: The Impact of Free Fatty Acid (FFA-) Suppression on Myocardial Lipids and Function in Patients With Type 2 Diabetes
Acronym: HYPOTESIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Krebs, Prof.MD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HYPOTESIS; 2013-002656-32 (EudraCT Number)
Record Dates: First submitted 2013-10-26; First posted 2013-11-11 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acipimox+ (Experimental): 250 mg at 0 and 180 minutes (one day)
  Interventions: Drug: acipimox
- Placebo (Placebo Comparator): 1 Tablet at 0 and 180 minutes (one day)
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: acipimox
  Arms: acipimox+
Drug: Placebo Oral Capsule
  Arms: Placebo

SUMMARY:
There is evidence that inhibition of FFA-release by acipimox is associated with a significant decrease in myocardial lipid content (MYCL) as well as the ejection fraction (as a marker of systolic left ventricular function) in healthy subjects, indicating, that the heart is dependent on a constant supply of free fatty acids in order to guarantee normal cardiac function, and it further indicates, that the heart is not able to cover its energy demand by switching to glucose oxidation.

Since that phenomenon, better known as "metabolic inflexibility" has been mainly described in patients with diabetes, we aim to investigate the impact of FFA-inhibition on MYCL and cardiac function in patients with overt type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* HbA1C >6%

Exclusion Criteria:

* Insulin therapy (except: BOT=basal supported oral therapy)
* Known heart disease including coronary artery disease, cardiomyopathy, history of cardiac surgery
* Known intolerance against niacins
* Known contra-indications against magnetic resonance (MR-) examinations

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Krebs, Prof.MD, Principal Investigator — Medical University of Vienna, Dept. of Internal Medicine III, Division of Endocrinology and Metabolism
Locations (1):
- Division of Endocrinology and Metabolism, Internal Medicine III, Medical University of Vienna, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Groups:
- Acipimox First: Participants received acipimox 250 mg at 0 and 180 minutes on the first study day; after a wash out period of at least 2 weeks a second study day followed where they received a placebo capsule at 0 and 180 minutes
- Placebo: Participants received a placebo capsule at 0 and 180 minutes on the first study day; after a wash out period of at least 2 weeks a second study day followed where they received a acipimox 250 mg at 0 and 180 minutes
Period: Study Day 1
Arm/Group | Acipimox First | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Washout (at Least 2 Weeks)
Arm/Group | Acipimox First | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Study Day 2
Arm/Group | Acipimox First | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: On study day 1 subjects received acipimox 250 mg or placebo at 0 and 180 minutes (randomized, controlled, single blinded); after a wash out period of at least two weeks on study day 2 i) subjects who received acipimox 250 mg on study day 1 were administered placebo at 0 and 180 minutes and ii) subjects who received placebo on study day 1 were administered acipimox 250 mg at 0 and 180 minutes (randomized, controlled, single blinded).
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  Austria | 8

OUTCOME MEASURES:

1. Primary Outcome: MYCL
Description: Intramyocardiocellular lipid content (MYCL) before and after administration of acipimox or placebo
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: percentage of water signal
Groups:
- Acipimox+: 250 mg at 0 and 180 minutes (one day)
  acipimox
- Placebo: 1 capsule at 0 and 180 minutes (one day)
  placebo
Arm/Group | Acipimox+ | Placebo
Number analyzed (Participants) | 8 | 8
percentage of water signal
  Baseline | 0.54 (0.1) | 0.44 (0.1)
  180 minutes after administration | 0.35 (0.2) | 0.36 (0.1)

2. Secondary Outcome: Ejection Fraction
Description: Left ventricular ejection fraction before and after administration of acipimox or placebo
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Acipimox+ | Placebo
Number analyzed (Participants) | 8 | 8
percentage
  Baseline | 76 (6) | 78 (8)
  180 minutes after administration | 69 (9) | 77 (7)

3. Other Pre Specified Outcome: Stroke Volume
Description: Stroke volume before and after administration of acipimox or placebo
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: ml/m2
Arm/Group | Acipimox+ | Placebo
Number analyzed (Participants) | 8 | 8
ml/m2
  baseline | 38 (10) | 36 (6)
  180 minutes after administration | 31 (8) | 36 (6)

ADVERSE EVENTS:
Groups:
- Acipimox-: 1 Tablet at 0 and 180 minutes (one day)
  acipimox
Arm/Group | Acipimox+ | Acipimox-
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes